CLINICAL TRIAL: NCT01589068
Title: Effects of Progesterone on IV Nicotine Induced Changes on BOLD fMRI Signal, Hormones and Subjective Ratings of Stimulant Drugs
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinical studies never started; funds never received.
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Scott Lukas, PI, Mclean Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2006-p-001985
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2013-01

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine; Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Male Smokers (Active Comparator)
  Interventions: Drug: Intravenous Nicotine; Drug: Progesterone
- Female Smokers (Follicular Phase) (Active Comparator)
  Interventions: Drug: Intravenous Nicotine; Drug: Progesterone
- Female Smokers (Luteal Phase) (Active Comparator)
  Interventions: Drug: Intravenous Nicotine; Drug: Progesterone

INTERVENTIONS:
Drug: Intravenous Nicotine — Subjects will be given an IV challenge dose of nicotine or placebo in a constant volume of 2 mL on any study day. The nicotine solution (1.0 mg/70kg or 1.5 mg/70kg or 2.0 mg/70kg) will be administered over 1 min. This rate of drug delivery (2 mL over one minute) has been safe in our IRB-approved studies of nicotine. Most investigators have administered nicotine over 10 seconds without any adverse reactions. We concur with the IRB recommendation that the lower doses (1.0 mg/70kg and 1.5 mg/70 kg) will be administered first and the higher dose (2.0 mg/70kg) will be administered last.
  Other Names: IV Nicotine
Drug: Progesterone — To stimulate the luteal phase of the menstrual cycle, Prometrium capsules containing 200 mg of micronized progesterone or placebo (lactose containing) capsules will be administered orally at 120 minutes before the injection of IV nicotine.

SUMMARY:
The proposed clinical studies will analyze the interactions between progesterone, nicotine, fMRI measures of patterns of brain activity, covariance with endocrine hormones, mood and cardiovascular measures. It is hypothesized that the administration of progesterone at a dose that mimics luteal phase levels in normal cycling women will diminish the positive subjective effects of nicotine, as has been consistently observed for cocaine. This novel approach could have direct implications for facilitating smoking cessation treatment in women of reproductive age

DETAILED DESCRIPTION:
These clinical studies will examine the effects of progesterone on the acute effects of IV nicotine and on patterns of brain activation in areas of the brain with high levels of nicotine receptors. This will be correlated with serum nicotine levels, nicotine-induced changes in subjective states, and endocrine measures of the HPA and HPG axes. The temporal covariance of progesterone's effects on serum nicotine levels and nicotine-induced changes in subjective states and cardiovascular measures will be analyzed.

The covariance between the effects of progesterone on nicotine-induced changes in BOLD fMRI, endocrine, subjective and cardiovascular effects and the temporal concordance with increases in serum nicotine and cotinine levels will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 40 who currently smoke at least 15 cigarettes every day, and who fulfill DSM-IV diagnostic criteria for nicotine dependence will be eligible for participation.
* No evidence of clinically significant disease based upon complete medical history and physical examination by a qualified physician.
* Absence of DSM-IV Axis I Disorders other than nicotine dependence (305.10) as measured by the Structured Clinical Interview (SCID).
* Routine laboratory blood tests including complete blood count, electrolytes, BUN and creatinine, liver function tests, hepatitis panel and urinalysis will be performed. Laboratory parameters must be within the normal range. HBsAg must be negative but subjects who have hepatitis serology consistent with previous exposure to Hepatitis A, Hepatitis B, or Hepatitis C, but who do not have clinical and biochemical evidence of acute infection, will be acceptable.
* Hematocrit levels ≥ 39% for males and ≥ 35% for females.
* Serum pregnancy test (hCG beta subunit) results must be negative within 24 hrs of the study day.
* Normal ECG.
* A Body Mass Index (BMI-ratio of weight (W) to height (H) squared; W/H2=kg/m2) of between 18 and 27 for women and 21 to 29 for men.
* Subjects must be able to read and understand instructions, as well as provide a valid informed consent.
* Individuals without hypersensitivity to peanuts or peanut oil.
* Participants without a current diagnosis of lactose intolerance. No evidence of clinically significant disease based upon complete medical history and physical examination by a qualified physician.

Exclusion Criteria:

* Participants with any lifetime DSM-IV Axis I disorder other than nicotine dependence.
* Participants with clinically significant medical disorders.
* Women who are pregnant as determined by laboratory testing for serum beta hCG.
* Women who use hormonal contraceptive medications will not be accepted, because this would confound the hormonal measures.
* Women with a mean BMI of outside the range 18-27 and men with a BMI outside the range 21-29.
* Participants who describe themselves as seeking treatment will not be selected but will be referred to local smoking cessation programs.
* Participants with allergies to peanuts or peanut oil.
* Participants diagnosed with lactose intolerance.
* Participants with ferromagnetic implants or other contraindications to fMRI:

  * Cardiac pacemakers
  * Metal clips on blood vessels (also called stents)
  * Artificial heart valves
  * Artificial arms, hands, legs, etc.
  * Brain stimulator devices
  * Implanted drug pumps
  * Ear implants
  * Eye implants or known metal fragments in eyes
  * Exposure to shrapnel or metal filings (wounded in military combat, sheet metal workers, welders, and others)
  * Other metallic surgical hardware in vital areas
  * Certain tattoos with metallic ink
  * Transdermal patches (eg. Orthro Evra, Nicoderm CQ)
  * Metal IUD (s)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Effect of progesterone on IV nicotine, hormones and subjective ratings | From baseline to study completion (approximately 8 months for males and 2 years for females)
  We are examining the effects of progesterone on the acute effects of IV nicotine and BOLD signal active in areas of the brain with high levels of nicotine receptors. Correlational analyses between brain activation patterns, serum nicotine levels, serum/plasma hormone levels, and nicotine-induced changes in subjective statues, as measured by a visual analog scale, are being evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy K Mello, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- Alcohol and Drug Abuse Research Center at McLean Hospital, Belmont, Massachusetts, United States